CLINICAL TRIAL: NCT00886574
Title: Multi-Center, Randomized, Open Label Study of the Efficacy of Cilostazol Versus Aspirin for Primary Prevention of Atherosclerotic Events With Korean Type 2 DM Patients
Brief Title: Cilostazol Versus Aspirin for Primary Prevention of Atherosclerotic Events
Acronym: CAPPA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanyang University (Other)
Collaborators: Ajou University School of Medicine (Other); Kyunghee University Medical Center (Other); Korea University Guro Hospital (Other); Inha University Hospital (Other); Inje University (Other); Hallym University Medical Center (Other)
Responsible Party: Yongsoo, Park, M. D., Department of Internal Medicine, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HY-2009-11
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Cilostazol versus Aspirin; Anti-PLT drug; Primary Prevention of Atherosclerotic Events; Type 2 DM; Intima media thickness (IMT)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): Aspirin 100 mg once a day
  Interventions: Drug: Aspirin
- Cilostazol (Active Comparator): Cilostazol 200 mg (50 mg 2T twice per day)
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 200 mg (50 mg 2T twice per day)
  Other Names: Pletaal
  Arms: Cilostazol
Drug: Aspirin — 100 mg once a day
  Arms: Aspirin

SUMMARY:
This multi-center, randomized controlled study aims to evaluate the efficacy of Cilostazol versus Aspirin for primary prevention of atherosclerotic events with Korean type 2 Diabetes Mellitus (DM) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus with high risk of macrovascular complications; high risk is one or more as follows:

   * Hypertension (≧ 140/90 or anti-hypertensive therapy)
   * Hypercholesterolemia (LDL-C > 130 mg/dL or anti-hyperlipidemic therapy)
   * TG > 200 mg/dL
   * Non proliferative retinopathy or macular edema
   * Microalbuminuria or macroalbuminuria
   * Smoker
2. Patients on no anti PLT drug history
3. Patients who are agree with this research

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Macrovascular complication history
3. Uncontrolled hypertension, unstable angina history
4. Congestive heart failure
5. Bleeding tendency
6. Chronic liver disease (ALT > 100 or AST > 100) or Chronic renal disease creatinine > 3.0 mg/dl)
7. Anemia (hemoglobin < 10 mg/dl) or thrombocytopenia (platelet count less than 100,000/mm3)
8. Pregnant or lactation women
9. Plan to be revascularized in 4 weeks
10. Plan to go to surgery or invasive intervention in 4 weeks
11. Plan to need to admission for acute cardiovascular disease in 4 weeks
12. Contraindication of this medication
13. Other anti-PLT drug therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Maximal and mean intima media thickness (IMT) of both common carotid artery of the cilostazol group in comparison with the aspirin group | every 6 months following randomization, for 48 months

SECONDARY OUTCOMES:
Events of the ischemic heart disease | every 12 months following randomization, for 48 months
Events of cerebrovascular disease | every 12 months following randomization, for 48 months
Events of peripheral vascular disease | every 12 months following randomization, for 48 months
Events of hemorrhagic vascular complication | every 12 months following randomization, for 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongsoo Park, M.D. Ph.D, Principal Investigator — Department of Internal Medicine, Hanyang University
Locations (6):
- South Korea (6):
  - Inha University Hospital, Incheon
  - Hallym University Hospital, Pyungcheon
  - Hallym University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung hee University Medical Center, Seoul
  - Ajou University Hospital, Suwon